CLINICAL TRIAL: NCT03441217
Title: Hyoscine Butylbromide Effect on Duration of Labor in Nulliparous Women: A Randomized, Double Blind, Controlled Trial
Brief Title: Hyoscine Butylbromide Effect on Duration of Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Thomas Hospital, Panama (Other)
Collaborators: Sistema Nacional de Investigadores de Panamá (Unknown)
Responsible Party: Principal Investigator, Osvaldo A. Reyes T., Head - Research Department, Saint Thomas Hospital, Panama
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MHST2014-05
Record Dates: First submitted 2018-02-13; First posted 2018-02-22 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Labor
Keywords: Duration of labor; Hyoscine butylbromide
MeSH Terms: interventions — Butylscopolammonium Bromide; Injections; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyoscine Butylbromide 20Mg/1mL Injection (Experimental): Nulliparous women with gestations at term receive 20 mg of Hyoscine butylbromide IV upon arrival in the Labor and Delivery Unit (4-5 cms).
  Interventions: Drug: Hyoscine Butylbromide 20Mg/1mL Injection
- Saline solution (Placebo Comparator): Nulliparous women with gestations at term receive Saline Solution IV upon arrival in the Labor and Delivery Unit (4-5 cms).
  Interventions: Drug: Saline Solution

INTERVENTIONS:
Drug: Hyoscine Butylbromide 20Mg/1mL Injection — Nulliparous women with gestations at term receive 20 mg of Hyoscine butylbromide upon arrival in the Labor and Delivery Unit (4-5 cms).
  Arms: Hyoscine Butylbromide 20Mg/1mL Injection
Drug: Saline Solution — Nulliparous women with gestations at term receive 20 mg of saline solution upon arrival in the Labor and Delivery Unit (4-5 cms).
  Arms: Saline solution

SUMMARY:
To evaluate the duration of labour (active phase of labour) in nulliparous women with gestations between 37 and 41 6/7 weeks when 20 mg of Hyoscine butylbromide was applied intravenously and compared with similar patients that received a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Low risk gestation between 37 and 41 6/7 weeks.
* Cephalic (vertex) presentation.
* Spontaneous labor in active phase (4 cms)

Exclusion Criteria:

* Premature rupture of membranes upon arrival at the Labor and Delivery Unit > 4 hours.
* Multiple order pregnancy.
* Stillbirth.
* Any fetal condition that could interfere in the mode of delivery (macrosomia, fetal growth restriction, oligohydramnios).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2019-07-12 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Duration of first stage of labor | 24 hours
  Time measured from the moment the patient receive the allocated medication/placebo to complete dilation
Rate of cervical dilation | 24 hours
  Speed of cervical dilation (cms/hour) from the moment the patient receive the allocated medication/placebo to complete dilation

SECONDARY OUTCOMES:
Duration of labor | 24 hours
  Time measured from the moment the patient receive the allocated medication/placebo to delivery
Fetal and neonatal complications | 72 hours
  Number of adverse events (fetal or neonatal)

CONTACTS AND LOCATIONS:
Overall Officials: Osvaldo Reyes, MD, Study Director — Maternidad del Hospital Santo Tomás
Locations (1):
- Saint Thomas Maternity Hospital, Panama City, Panama

IPD SHARING:
Plan to Share IPD: No